CLINICAL TRIAL: NCT00383552
Title: A 26-Week Placebo-Controlled Efficacy and Safety Study of Mometasone Furoate/Formoterol Fumarate Combination Formulation Compared With Mometasone Furoate and Formoterol Monotherapy in Subjects With Persistent Asthma Previously Treated With Low-Dose Inhaled Glucocorticosteroids
Brief Title: Effects of Mometasone Furoate/Formoterol Combination Versus Mometasone Furoate Alone in Persistent Asthmatics (Study P04073AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04073; Doc ID: 3100873;; EUDRACT No: 2006-001577-13;
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; BID protein, human; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MF/F MDI 100/10 mcg BID (Experimental)
  Interventions: Drug: Mometasone Furoate/Formoterol Fumarate Combination MDI 100/10 mcg BID
- MF MDI 100 mcg BID (Experimental)
  Interventions: Drug: Mometasone Furoate MDI (MF MDI)
- F MDI 10 mcg BID (Experimental)
  Interventions: Drug: Formoterol Fumarate 10 mcg
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate/Formoterol Fumarate Combination MDI 100/10 mcg BID — MF/F 100/10 mcg via a metered dose inhaler (MDI) twice daily for 26 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 100/10 mcg BID
Drug: Mometasone Furoate MDI (MF MDI) — MF 100 mcg via metered dose inhaler twice daily for 26 weeks
  Other Names: SCH 32088
  Arms: MF MDI 100 mcg BID
Drug: Formoterol Fumarate 10 mcg — F via metered dose inhaler 10 mcg twice a day for 26 weeks
  Other Names: Foradil
  Arms: F MDI 10 mcg BID
Drug: Placebo — Placebo metered dose inhaler twice a day for 26 weeks
  Arms: Placebo BID

SUMMARY:
This is a randomized, multi-center, double-blind, double-dummy, placebo-controlled, parallel-group study, evaluating the efficacy of mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) versus MF for 26 weeks. Prior to the 26-week double-blind Treatment Period, participants will receive open-label (OL) MF MDI 100 mcg twice daily (BID) for 2 to 3 weeks during the Run-in Period. Efficacy will be measured by the Area Under the Curve from 0 to 12 hours [AUC](0-12 hours) of the change from Baseline to the Week 12 Endpoint in Forced Expiratory Volume in One Second (FEV1) and by the time-to-first severe asthma exacerbation across the 26-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* >=12 years, either sex, any race, asthma diagnosis >=12 months that is consistent with the following: Diagnosis based on clinical history & examination, pulmonary function parameters & response to beta-2-agonists, according to international guidelines.
* Been using low daily dose of inhaled corticosteroid (ICS) (either alone or in combination with long-acting beta agonist [LABA]) >=12 weeks & been on stable asthma regimen for >=2 weeks prior to Screening. Low daily doses of ICS are:

200-500 mcg beclomethasone chlorofluorocarbon (CFC),

100-250 mcg beclomethasone hydrofluoroalkane (HFA),

200-600 mcg budesonide dry powder inhaler (DPI),

500-1000 mcg flunisolide,

100-250 mcg fluticasone,

200 mcg MF,

400-1000 mcg triamcinolone acetonide,

80 to 160 mcg ciclesonide.

Note: Dose delivery by method/modality other than these must be equivalent.

* No harm in changing current asthma therapy to investigator, subject (legal representation, if applicable) must be willing to discontinue his/her ICS or ICS/LABA combination prior to initiating MF MDI run-in medication at Screening Visit, & transferred to open-label treatment with MF MDI 100 mcg BID for 2-3 weeks prior to Baseline Visit.
* To document diagnosis of asthma & assure responsiveness to bronchodilators before randomization 1 of these can be used at Screening Visit or thereafter, but prior to Baseline Visit:

Demonstrate increase in absolute FEV1 >=12% & >=200 mL within approximately 15 to 20 minutes after administration of 4 inhalations of albuterol/salbutamol (total dose 360-400 mcg) or nebulized short-acting beta agonist (SABA) (2.5 mg) if confirmed as standard office practice, OR

Demonstrate peak expiratory flow (PEF) variability >20% expressed as percentage of the mean highest & lowest morning prebronchodilator (before taking albuterol/salbutamol) PEF over >=1 week, OR

Demonstrate diurnal variation in PEF of >20% based on difference between prebronchodilator (before taking albuterol/salbutamol) morning value & postbronchodilator value (after taking albuterol/salbutamol) from evening before, expressed as percentage of mean daily PEF value.

* At Screening Visit, FEV1 must be >=60% & <=90% predicted.
* At Baseline Visit, FEV1 must be >=60% & <=85% predicted when all restricted drugs have been withheld for appropriate intervals.
* Lab tests at Screening Visit must be normal or acceptable to investigator/sponsor and include serum pregnancy for females of child-bearing potential). Electrocardiogram (ECG) at Screening Visit, using centralized trans-telephonic technology must be acceptable to investigator. Chest x-ray performed at Screening Visit or within 12 months prior to Screening Visit must be acceptable to investigator.
* Subject (legal representation, if applicable) must be willing to give written informed consent & able to adhere to schedules.
* A non-pregnant woman of childbearing potential must use birth control. Includes: hormonal contraceptives including hormonal vaginal ring, hormonal implant or depot-injectable; Intrauterine device (IUD); medically prescribed topically-applied transdermal contraceptive patch; condom in combination with spermicide; monogamous relationship with male who had vasectomy. Started birth control method >=3 months prior to Screening (exception condom), & must agree to continue its use. Female of childbearing potential who is not currently sexually active must agree & consent to using birth control, should she become active. Women who have been surgically sterilized or are >=1 year postmenopausal are not considered to be of childbearing potential. Female must have negative serum pregnancy test at Screening.

Exclusion Criteria:

* Increase/decrease in absolute FEV1 of >20% at any time from Screening Visit up to & including Baseline Visit. Pulmonary function tests (PFTs) will be performed in the morning.
* >8 inhalations/day of SABA MDI or >=2 nebulized treatments/day of 2.5 mg SABA on 2 consecutive days from Screening Visit up to & including Baseline Visit.
* Decrease in AM/PM PEF below Screening Period stability limit on 2 consecutive days prior to randomization.
* Asthma deterioration results in emergency treatment, hospitalization, or treatment with additional, excluded asthma medication (including oral or other systemic corticosteroids, but allowing SABA) as judged by investigator at any time from Screening Visit up to & including Baseline Visit.
* Treated in emergency room (ER) (for severe asthma exacerbation requiring systemic glucocorticosteroid treatment) or admitted to hospital for management of airway obstruction within last 3 months.
* Ever required ventilator support for respiratory failure secondary to asthma.
* Upper/lower respiratory tract infection within previous 2 weeks prior to Screening & Baseline Visits. Visits can be rescheduled 2 weeks after complete resolution.
* Smoker or ex-smoker & has smoked within previous year or has cumulative smoking history >10 pack-years.
* Significant abnormal vital sign.
* Evidence upon visual inspection of significant oropharyngeal candidiasis at Baseline or earlier with or without treatment. If there is evidence at Screening or Pre-Baseline Visit, may be treated as appropriate & Baseline Visit can be scheduled upon resolution.
* History of significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular, or other which, in judgment of investigator, could interfere with study or require treatment which might interfere with study. Examples include (but are not limited to) insulin-dependent diabetes, hypertension being treated with beta-blockers, active hepatitis, coronary artery disease, arrhythmia, significant QTc prolongation (ie QTcF or QTcB [Fridericia or Bazett corrections, respectively >500 msecs), stroke, severe rheumatoid arthritis, chronic open-angle glaucoma or posterior subcapsular cataracts (including prior cataract surgery), acquired immune deficiency syndrome (AIDS), or conditions that may interfere with respiratory function such as chronic obstructive pulmonary disease (COPD), chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis. Others which are well-controlled & stable (eg hypertension not requiring beta-blockers) will not prohibit participation if deemed appropriate by investigator.
* Allergic/intolerant of glucocorticoids, beta-2-agonists, or any inactive excipients in study drugs.
* Female who is breast-feeding, pregnant, or intends to become pregnant while in study.
* Illicit drug user.
* Human immunodeficiency virus (HIV) positive (testing not done).
* Unable to use oral MDI inhaler.
* Has been taking any restricted medications prior to Screening without meeting required washout.
* Cannot adhere to prohibited & permitted concomitant medications.
* May not participate in same study at another site. Cannot participate in different study at any site, during same time.
* Must not be randomized into study more than once.
* No person directly associated with administration of study may participate.
* Previously participated in trial with MF/F.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meltzer EO, Kuna P, Nolte H, Nayak AS, Laforce C; P04073 Study Investigators. Mometasone furoate/formoterol reduces asthma deteriorations and improves lung function. Eur Respir J. 2012 Feb;39(2):279-89. doi: 10.1183/09031936.00020310. Epub 2011 Aug 4. PMID 21828036

RESULTS

PARTICIPANT FLOW:
Groups:
- MF/F MDI 100/10 mcg BID: Mometasone Furoate/Formoterol Fumarate (MF/F) metered dose inhaler (MDI) 100/10 mcg twice daily (BID)
- MF MDI 100 mcg BID: Mometasone Furoate (MF) metered dose inhaler (MDI) 100 mcg twice daily (BID)
- F MDI 10 mcg BID: Formoterol Fumarate (F) metered dose inhaler (MDI) 10 mcg twice daily (BID)
- Placebo BID: Placebo twice daily (BID)
Period: Overall Study
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Started | 182 | 188 | 188 | 188
Completed | 146 | 147 | 127 | 116
Not Completed | 36 | 41 | 61 | 72
Not completed — Adverse Event | 7 | 6 | 9 | 6
Not completed — Lack of Efficacy | 4 | 13 | 29 | 42
Not completed — Lost to Follow-up | 0 | 1 | 5 | 1
Not completed — Did not wish to continue (unrelated) | 4 | 9 | 5 | 6
Not completed — Did not wish to continue (related) | 1 | 0 | 2 | 3
Not completed — Noncompliance with the protocol | 11 | 6 | 8 | 10
Not completed — Did not meet protocol eligibility | 8 | 6 | 2 | 3
Not completed — Administrative | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID | Total
Number analyzed (Participants) | 182 | 188 | 188 | 188 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (16.9) | 39.4 (16.7) | 38.5 (15.6) | 38.1 (17.4) | 38.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 105 | 103 | 106 | 413
  Male | 83 | 83 | 85 | 82 | 333

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Time Curve From 0 to 12 Hours (AUC(0-12 Hours)) of Change From Baseline to Week 12 in Forced Expiratory Volume (Liters) in 1 Second (FEV1)
Description: The average of the two predose FEV1 measurements (30 minutes prior to dosing and 0 hour, immediately prior to dosing) at the Baseline Visit were subtracted from each of the serial measurements over the 12-hour period. The AUC was calculated based on these changes from Baseline evaluations. The comparison was for MF/F vs MF. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: Efficacy analyses were based on randomized participants with Baseline and any post-baseline data (intent-to-treat principle).
Measure: Least Squares Mean (Standard Deviation); unit: liters * hours
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 155 | 156 | 146 | 129
liters * hours
  Baseline | 3.94 (3.29) | 1.85 (3.29) | 4.09 (3.29) | 1.64 (3.29)
  Change from Baseline | 4.00 (3.71) | 2.53 (3.71) | 3.83 (3.71) | 1.11 (3.71)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs MF MDI 100 mcg BID; Test type: Superiority or Other; p = 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline to Week 26 in the Asthma Control Questionnaire (ACQ) Total Score
Description: ACQ consists of seven questions each scaled from 0 (best case) to 6 (worst case). The comparison was for MF/F vs placebo. Standard deviation was pooled.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 143 | 145 | 129 | 116
units on a scale
  Baseline | 1.34 (0.71) | 1.29 (0.60) | 1.38 (0.76) | 1.23 (0.71)
  Change from Baseline | -0.40 (0.65) | -0.32 (0.65) | -0.12 (0.65) | -0.11 (0.65)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.001, ANCOVA

3. Primary Outcome: Median Time-to-first Severe Asthma Exacerbation Over the 26-week Treatment Period
Description: Severe asthma exacerbation refers to an occurrence of a decrease below 80% of Baseline in FEV1, a decrease below 70% of Baseline in PEF on 2 consecutive days or a clinical deterioration of asthma resulting in emergency treatment, hospitalization or treatment with asthma medication.
Time Frame: Across the 26 week treatment period
Population: Medians for time-to-event outcomes are estimated for those who had events.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MF/F MDI 100/10 Mcg BID | MF MDI 100 Mcg BID | F MDI 10 Mcg BID | Placebo BID
Number analyzed (Participants) | 30 | 53 | 84 | 86
Days | 45.5 (101) [11 to 101] | 54 (98) [12 to 98] | 51.5 (125.5) [16.5 to 125.5] | 27.5 (87) [8 to 87]

4. Secondary Outcome: Change From Baseline to Week 26 in Asthma Quality of Life Questionnaire With Standarized Activities (AQLQ[S]) Total Score
Description: AQLQ(S) consists of 32 questions each scaled from 1 (worst case) to 7 (best case). The comparison was for MF/F vs placebo. Standard deviation was pooled.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 144 | 147 | 129 | 117
units on a scale
  Baseline | 5.60 (0.93) | 5.65 (1.00) | 5.60 (0.98) | 5.76 (1.02)
  Change from Baseline | 0.44 (0.73) | 0.39 (0.73) | 0.15 (0.73) | 0.06 (0.73)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Change From Baseline in Proportion of Nights Across the Treatment Period With Nocturnal Awakenings Due to Asthma Which Require Use of Short-acting Beta Agonists (SABA)
Description: Baseline is the proportion of nights of the last week (Days -7 to 1) prior to first dose with nocturnal awakenings. Scale is measured as 0 to 1 with 0=no awakenings to 1=awakenings every night. The comparison was for MF/F vs placebo. Standard deviation was pooled.
Time Frame: Baseline to Endpoint
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Proportion of Nights
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 181 | 185 | 185 | 188
Proportion of Nights
  Baseline | 0.13 (0.12) | 0.12 (0.12) | 0.15 (0.15) | 0.13 (0.14)
  Change from Baseline | -0.06 (0.16) | -0.03 (0.16) | -0.03 (0.16) | 0.02 (0.16)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change From Baseline in AM FEV1 Pre-dose Assessment, or Trough FEV1, at Week 12
Description: Trough FEV1 is a measure of the end-of-dosing interval. The comparison was for MF/F vs F. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: liters
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 160 | 163 | 160 | 137
liters
  Baseline | 2.50 (2.56) | 2.41 (2.46) | 2.47 (2.52) | 2.46 (2.50)
  Change from Baseline | 0.18 (0.21) | 0.16 (0.21) | 0.11 (0.21) | 0.04 (0.21)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p = 0.073, Longitudinal Model

7. Secondary Outcome: AUC(0-12 Hour) of the Change From Baseline to Week 12 in FEV1 for Each Body Mass Index (BMI) Subgroup
Description: The average of the two predose FEV1 measurements (30 minutes prior to dosing and 0 hour, immediately prior to dosing) at the Baseline Visit were subtracted from each of the serial measurements over the 12-hour period. The AUC was calculated based on these changes from Baseline evaluations. BMI is a number calculated from a person's weight and height. The higher the number, the higher the amount of fat. The comparison was for MF/F vs placebo. Standard deviation was pooled.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: liters * hours
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 155 | 156 | 146 | 128
liters * hours
  Less than 25 | 5.24 (4.42) | 3.19 (4.42) | 4.34 (4.42) | 2.22 (4.42)
  25 to less than 30 | 3.36 (4.14) | 3.23 (4.14) | 4.26 (4.14) | 1.22 (4.14)
  30 or more | 3.35 (3.68) | 1.69 (3.68) | 3.13 (3.68) | -0.73 (3.68)
Statistical Analysis 1: Comparison: MF/F MDI 100/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p = 0.015, ANCOVA — BMI 25 to <30
Statistical Analysis 2: Comparison: MF/F MDI 100/10 mcg BID vs Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA — BMI less than 25 and for BMI 30 or more

8. Primary Outcome: Number of Participants With at Least One Severe Asthma Exacerbation at Week 26
Description: Severe asthma exacerbation refers to an occurrence of a decrease below 80% of Baseline in FEV1, a decrease below 70% of Baseline in PEF on 2 consecutive days and or a clinical deterioration of asthma resulting in emergency treatment, hospitalization or treatment with asthma medication.
Time Frame: Week 26
Measure: Number; unit: participants
Arm/Group | MF/F MDI 100/10 mcg BID | MF MDI 100 mcg BID | F MDI 10 mcg BID | Placebo BID
Number analyzed (Participants) | 155 | 156 | 146 | 129
participants | 30 | 53 | 84 | 86

ADVERSE EVENTS:
Description: All participants treated with OL MF MDI and/or double-blind study medication are included in the safety population.
Groups:
- OL MF MDI 100 MCG BID: Open-label (OL) mometasone furoate (MF) metered dose inhaler (MDI) 100 mcg twice daily (BID). Participants received 2- to 3-weeks (approximately) of open-label run-in with MF MDI 100 mcg BID prior to the 26-week double-blind Treatment Period.
Arm/Group | OL MF MDI 100 MCG BID | MF/F MDI 100/10 MCG BID | MF MDI 100 MCG BID | F MDI 10 MCG BID | PLACEBO
Serious Adverse Events (participants affected / at risk) | 2/882 | 4/182 | 5/188 | 1/188 | 1/188
Other Adverse Events (participants affected / at risk) | 22/882 | 33/182 | 37/188 | 32/188 | 24/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL MF MDI 100 MCG BID (N=882) | MF/F MDI 100/10 MCG BID (N=182) | MF MDI 100 MCG BID (N=188) | F MDI 10 MCG BID (N=188) | PLACEBO (N=188)
PULMONARY VALVE STENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GOITRE (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL PERICARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL MF MDI 100 MCG BID (N=882) | MF/F MDI 100/10 MCG BID (N=182) | MF MDI 100 MCG BID (N=188) | F MDI 10 MCG BID (N=188) | PLACEBO (N=188)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 17 (19) | 13 (15) | 7 (7) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 10 (11) | 17 (19) | 20 (26) | 12 (17)
HEADACHE (Nervous system disorders) | 15 (18) | 12 (17) | 11 (18) | 9 (9) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results without prior

sponsor written consent. The investigator agrees to provide to the sponsor, 45 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues/disagreement.